CLINICAL TRIAL: NCT05160779
Title: Impact of Genetic Polymorphisms of Vasoactive Peptides on the Prognosis of Patients Diagnosed With Mild and Severe Cases of COVID19
Brief Title: Impact of Genetic Polymorphisms of Vasoactive Peptides on the Prognosis of Patients With COVID19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leonardo Paroche de Matos (Other)
Collaborators: Prof. Dr. José Antônio Silva Júnior (Unknown); Msc. Allan Luis Barboza Atum (Unknown)
Responsible Party: Principal Investigator, Leonardo Paroche de Matos, Msc; Doctoral student in medicine at the Universidade Nove de Julho, Leonardo Paroche de Matos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20211214
Record Dates: First submitted 2021-12-14; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Sars-CoV-2 Infection
Keywords: SARS-CoV-2 infection; Genetic polymorphism; Polymerase Chain Reaction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The allocation of participants in the two research groups will happen in a stratified random way, so that individuals who were diagnosed and presented the mild or asymptomatic form of the disease (with treatment and monitoring carried out by primary care) will be gathered in the study group called " mild/asymptomatic cases", and individuals who were diagnosed and presented with severe forms of the disease, and who required hospitalization in the Intensive Care Unit (ICU) (with or without invasive mechanical ventilation) will be grouped in the group called "severe cases ".
Masking Description: No masking of groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild/asymptomatic cases (Active Comparator): For the collection of cells from the oral cavity, a sterile swab will be used for the procedure, and will be opened by the collector in the presence of the participant. The biological material will be collected from the participant's cheek mucosa (rotating the swab 360º using light pressure (approximately 75N) on the mucosa tissue and then packed in a tube containing 3ml of sterile 0.9% saline solution) of the participant. confirmation of identification data in order to analyze and relate polymorphisms found in components of vasoactive peptide systems in DNA samples collected from patients diagnosed with SARS-CoV-2 (COVID-19) who developed mild or asymptomatic conditions.
  Interventions: Other: Analysis of genetic polymorphisms of vasoactive peptides in COVID-19
- Serious cases (Active Comparator): For the collection of cells from the oral cavity, a sterile swab will be used for the procedure, and will be opened by the collector in the presence of the participant. The biological material will be collected from the participant's cheek mucosa (rotating the swab 360º using light pressure (approximately 75N) on the mucosa tissue and then packed in a tube containing 3ml of sterile 0.9% saline solution) of the participant. confirmation of identification data in order to analyze and relate polymorphisms found in components of vasoactive peptide systems in DNA samples collected from patients diagnosed with SARS-CoV-2 (COVID-19) who developed severe pathology.
  Interventions: Other: Analysis of genetic polymorphisms of vasoactive peptides in COVID-19

INTERVENTIONS:
Other: Analysis of genetic polymorphisms of vasoactive peptides in COVID-19 — Evaluate the frequency of the insertion/deletion (I/D) polymorphism in the ACE gene; to assess the frequency of polymorphism in the bradykinin B2 receptor gene; to assess the frequency of the polymorphism in the CK-M gene and compare the frequencies of these polymorphisms between patients with severe and mild conditions.

SUMMARY:
Introduction: A pandemic such as the SRAS-CoV-2 (COVID-19) has a great negative socioeconomic impact with very limited therapeutic options. As with any disease, a detailed understanding of its pathophysiological mechanisms is critical for the development of new therapies. In SRAS-CoV-2, few studies have verified a possible relationship of these vasoactive peptide polymorphisms with patient prognosis. Objective: To analyze and relate polymorphisms found in components of vasoactive peptide systems in DNA samples collected from patients diagnosed with SARS-CoV-2 (COVID-19) who developed severe conditions and patients infected with mild or asymptomatic conditions. Methodology: Cross-sectional, analytical and qualitative study that will be conducted with approximately 151 participants previously diagnosed with SARS-CoV-2 with mild or asymptomatic forms of the pathology, diagnosed in primary care in the city of Guarulhos/SP- specifically in the Basic Health Unit of Nova Saúde Bonsucesso- well with participants who were diagnosed with the severe forms that required hospitalization in 2021. For the collection of biological material, a sterile swab will be used in order to collect cells from the oral cavity, specifically from the oral mucosa. Expected results: We hope to identify and relate the polymorphisms of vasoactive peptide genes from patients with mild, asymptomatic or severe forms of SARS-CoV-2 infection, thus contributing to the understanding of the different clinical evolutions of the disease.

DETAILED DESCRIPTION:
Cross-sectional, analytical and qualitative study that will be carried out with approximately 151 participants who were previously diagnosed with SARS-CoV-2 with mild and severe symptoms of the pathology, diagnosed in primary care in the city of Guarulhos/SP - specifically in the Basic Health Unit Nova Bonsucesso or who have a history of previous admissions - requiring hospitalization in the year 2021 (which will be removed from the COVID case monitoring spreadsheet available at the study UBS). Cells will be collected from the participants' oral cavity using a sterile cotton swab. The collections will be carried out at the Basic Health Unit Nova Bonsucesso, located in the city of Guarulhos/SP (mild/asymptomatic cases), under the supervision and responsibility of the dentist and collaborator of this Leonardo Paroche de Matos project. The Free and Informed Consent Form will be filled out and signed after guidance on the research and its subsequent acceptance by the participant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years old
* With or without associated comorbidities: any pathology of the systems: cardiovascular, respiratory, endocrine, digestive, neurological, psychiatric, genitourinary
* Diagnosed with COVID-19 through RT-PCR (naso-oropharyngeal swab)
* Who agreed to participate in the research voluntarily

Exclusion Criteria:

* Participants who refuse to participate in the survey
* Who have lesions in the oral mucosa that make the collection of material unfeasible
* Individuals with severe xerostomia
* In cancer treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between polymorphisms and COVID-19 progression | 1 month
  To investigate a possible correlation between gene polymorphism and disease progression (SARS-CoV-2) for asymptomatic, mild or severe conditions

CONTACTS AND LOCATIONS:
Overall Officials: José Antônio Silva Júnior, PhD, Study Director — University Ninth of July
Locations (2):
- Brazil (2):
  - Guarulhos City Hall, Guarulhos, São Paulo
  - University Ninth of July, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared at any stage of the survey.